CLINICAL TRIAL: NCT00312351
Title: An Exploratory Randomized, Double-Masked, Multi-Center Comparative Trial, in Parallel Groups, to Explore the Safety and Efficacy of Three Different Doses of Intravitreous Injections of Pegaptanib Sodium (Anti-VEGF Pegylated Aptamer) Given Every 6 Weeks for 102 Weeks, in Patients With Subfoveal Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: A Clinical Trial to Explore the Safety and Efficacy of Three Different Doses of Pegaptanib Sodium in Patients With Wet Age-Related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOP1014
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Macular Degeneration
Keywords: AMD; Age-Related Macular Degeneration; Macular Degeneration; Macugen; pegaptanib sodium; ERG; specular microscopy; Age-Related Mcular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

INTERVENTIONS:
Drug: Pegaptanib sodium

SUMMARY:
The purpose of this trial is to compare the ability of three different doses of pegaptanib sodium to safely and effectively minimize fluid leakage within the eye, thereby stabilizing or improving vision in patients with wet AMD. The study will also examine the effects of pegaptanib sodium on the cornea and sensory retina of patients with wet AMD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender, aged 50 years or greater.
* Subfoveal choroidal neovascularization (CNV) due to AMD.
* Best corrected visual acuity in the study eye between 20/40 and 20/320.
* Normal electroretinogram, and corneal endothelial cell density of 1500 cells/mm2 or more.

Exclusion Criteria:

* Any prior photodynamic therapy (PDT) with Visudyne or thermal laser to the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262
Dates: Start 2006-04; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Locations (1):
- Charlotte Eye, Ear, Nose and Throat Associates, P.A., Charlotte, North Carolina, United States